CLINICAL TRIAL: NCT04123392
Title: Decitabine+Busulfan+Cyclophosphamide vs Busulfan+Cyclophosphamide Conditioning Regimen for TP53+ Myeloid Tumors Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Decitabine + BUCY vs BUCY Conditioning Regimen for TP53+ Myeloid Tumors Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP53+ Myeloid tumors
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: TP53; Myeloid Tumors; Conditioning; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Decitabine; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine + BUCY (Experimental): For TP53+ myeloid tumors undergoing allo-HSCT, Decitabine +BUCY conditioning regimen was Decitabine 20mg/m2/day on days -14 and -10, Busulfan (BU) 3.2 mg/kg/day on days -7 and -4, Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Decitabine; Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)
- BUCY (Active Comparator): For TP53+ myeloid tumors undergoing allo-HSCT, BUCY conditioning regimen was Busulfan (BU) 3.2 mg/kg/day on days -7 and -4, Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Decitabine — Decitabine was administered at 20mg/m2/day on days -14 and -10.
  Arms: Decitabine + BUCY
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.

SUMMARY:
Recent studies have demonstrated that allogeneic hematopoietic stem cell transplantation (allo-HSCT) could be a valuable treatment choice for TP53+ myeloid tumors, such as acute myeloid leukemia and myelodysplastic syndrome. Unfortunately, some patients relapsed after allo-HSCT. In this prospective randomized controlled study, the safety and efficacy of Decitabine + BUCY and BUCY myeloablative conditioning regimens in TP53+ myeloid tumors undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Recent studies have demonstrated that allogeneic hematopoietic stem cell transplantation (allo-HSCT) could be a valuable treatment choice for TP53+ myeloid tumors, such as acute myeloid leukemia and myelodysplastic syndrome. BUCY conditioning regimen is the standard myeloablative regimen for TP53+ myeloid tumors undergoing allo-HSCT. However, it appears to have higher relapse rate and lower survival. To reduce the relapse rate and improve the survival, decitabine is added in the conditioning regimen. In this prospective randomized controlled study, the safety and efficacy of Decitabine + BUCY and BUCY myeloablative conditioning regimens in TP53+ myeloid tumors undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* TP53+ Myeloid tumors undergoing allo-HSCT
* 14-65 years

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
relapse rate | 1 year
  relapse rate

SECONDARY OUTCOMES:
overall survival (OS) | 1 year
  overall survival (OS)
disease-free survival (DFS) | 1 year
  disease-free survival (DFS)
transplant-related mortality (TRM) | 1 year
  transplant-related mortality (TRM)

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China